CLINICAL TRIAL: NCT02293512
Title: A Comparison of CBT and CET Interventions for Veterans With Tinnitus
Brief Title: A Comparison of Three Psychoeducational Group Interventions for Veterans With Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C1578-P; RX001578 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2014-11-05; First posted 2014-11-18 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Tinnitus
Keywords: Tinnitus; Coping; Psychoeducational intervention
MeSH Terms: conditions — Tinnitus | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Coping Effectiveness Training (Experimental): Coping Effectiveness Training (CET) is provided in a 3-session intervention to facilitate coping strategies among individuals with tinnitus. The CET psychoeducational intervention teaches coping skills to increase understanding of stress and coping with tinnitus, and to help individuals better know how to match appropriate coping strategies, based on whether the stressful situation is changeable or not.
  Interventions: Behavioral: Coping Effectiveness Training
- Cognitive-behavioral therapy (Active Comparator): Cognitive-behavioral therapy (CBT) is provided in a 3-session psychoeducational intervention to reduce negative affectivity triggered by tinnitus. CBT treatments for tinnitus target the reduction of psychopathology by altering cognitive distortions, automatic thoughts, and core beliefs, as well as behavioral techniques to reduce physiological arousal.
  Interventions: Behavioral: Cognitive-behavioral therapy
- Acceptance and Commitment Therapy (Active Comparator): Acceptance and Commitment Therapy (ACT) is provided in a 3-session psychoeducational intervention to decrease resistance to tinnitus and increase committed action based on values, despite having tinnitus.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Wait-list control group (No Intervention): Wait-list control group involves no intervention. This is a 'usual care' group.

INTERVENTIONS:
Behavioral: Coping Effectiveness Training — A CET psychoeducational intervention is provided to increase understanding of stress and coping with tinnitus, and to better learn how to match appropriate coping strategies, based on whether the stressful situation is changeable or not.
  Other Names: CET
  Arms: Coping Effectiveness Training
Behavioral: Cognitive-behavioral therapy — CBT treatments for tinnitus target the reduction of psychopathology by altering cognitive distortions, automatic thoughts, and core beliefs, as well as behavioral techniques to reduce physiological arousal.
  Other Names: CBT
  Arms: Cognitive-behavioral therapy
Behavioral: Acceptance and Commitment Therapy — An ACT psycho-educational intervention to reduce distress and resistance about having tinnitus and to increase committed actions based on one's values.
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy

SUMMARY:
Tinnitus (i.e., ringing in the ears) is currently the most prevalent disability among Veterans. A range of clinical interventions has been created to systematically address the range of issues caused by tinnitus. While numerous interventions purport to promote coping strategies for tinnitus-related problems, few studies directly target and measure coping outcomes. The present pilot study proposes a comparison of coping outcomes after 3 psycho-educational groups: a cognitive-behavioral therapy (CBT) intervention, a Coping Effectiveness Training (CET) intervention, or an Acceptance and Commitment Therapy intervention among Veterans with tinnitus. These groups will be compared to a usual care group among Veterans and civilians with tinnitus. The proposed study will be the first application of CET to tinnitus. The primary goals of this study are to develop a CET protocol for tinnitus and to evaluate the effectiveness of CBT, CET, and ACT interventions to a usual care group. The long-term goal of this study is to improve the quality of life among individuals with tinnitus.

DETAILED DESCRIPTION:
Tinnitus (i.e., ringing in the ears) is currently the most prevalent disability in the VA system. Numerous clinical interventions have been created to systematically address the range of issues caused by tinnitus. Only a few tinnitus interventions have focused on coping strategies. Coping strategies are cognitive, affective, and behavioral attempts to master new events, such as the onset of a disability or an impairment like tinnitus, that are overwhelming to an individual, and that because of their newness, an individual does not necessarily have automatic, adaptive responses. Evidence suggests that CET is effective in facilitating adaptive coping strategies among individuals with several types of impairments or disabilities. The proposed study will be the first application of CET to a tinnitus population.

The present study proposes a development of a CET protocol for tinnitus and a pilot study that assesses the effectiveness of the CET and ACT interventions compared to the current clinical practice of using a CBT intervention. All 3 psycho-educational interventions will be compared to a usual care group. The overarching goal of the proposed pilot study is to gain information that can be used to provide individuals with tinnitus with the best care for helping them to more successfully cope with tinnitus.

The aims of this research are to: 1) develop a CET protocol for tinnitus by means of information gathered from two focus groups and from CET consultants; 2) to examine whether a 3-session CET psycho-educational intervention is more effective than a 3-session CBT psycho-educational intervention or a 3-session ACT psycho-educational intervention, as compared to a usual care, in increasing coping strategies among individuals with tinnitus.

ELIGIBILITY:
Inclusion Criteria:

Development Phase (Phase 1)-focus groups:

Inclusion criteria are the following (more details are provided below):

* 1) Veterans;
* 2) have chronic tinnitus that is sufficiently bothersome to warrant intervention-see below for explanation;
* 3) able to communicate in English;
* 4) willing and able to give written informed consent;
* 5) use hearing aids if needed; and
* 6) have participated in the PTM program at the VA Portland Healthcare System.

Testing Phase (Phase 2)-interventions:

Inclusion criteria are the following:

* 1) Veterans and civilians;
* 2) have a score of at least 25 on the Tinnitus Functional Index ([TFI]; Meikle, J.A. Henry, et al., 2012);
* 3) have two errors or less on a six-item cognitive screening instrument (Callahan, Unverzagt, Hui, Perkins, & Hendrie, 2002);
* 4) able to communicate in English;
* 5) willing and able to give written informed consent; and
* 6) use hearing aids if needed.

Exclusion Criteria:

Development Phase (Phase 1)-focus groups:

Exclusion criteria are:

* Not meeting inclusion criteria 1-6,
* nor have any other factor that would preclude full participation in the study.

Testing Phase (Phase 2)-interventions:

Exclusion criteria are:

* Not meeting inclusion criteria 1-6,
* having participated in the PTM program or Phase 1 of this study,
* or having any other factor that would preclude full participation in the study. Recruitment for Phase 2 will begin in year 1 once the CET protocol is finalized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin C Martz, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: VAPORHCS National Center for Rehabilitative Auditory Research (NCRAR) — http://www.ncrar.research.va.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Coping Effectiveness Training (CET): A 3-session intervention to facilitate coping strategies among individuals with tinnitus.
  Coping Effectiveness Training for tinnitus: A CET psycho-educational intervention to increase understanding of stress and coping with tinnitus, and to better learn how to match appropriate coping strategies, based on whether the stressful situation is changeable or not.
- Cognitive-behavioral Therapy (CBT): A 3-session intervention to reduce negative affectivity triggered by tinnitus.
  Cognitive-behavioral therapy (CBT): CBT treatments for tinnitus target the reduction of psychopathology by altering cognitive distortions, automatic thoughts, and core beliefs, as well as behavioral techniques to reduce physiological arousal.
- Acceptance and Commitment Therapy: A 3-session intervention to decrease resistance to tinnitus and increase committed action based on values, despite having tinnitus.
  Acceptance and Commitment Therapy for tinnitus: An ACT psycho-educational intervention to reduce distress and resistance about having tinnitus and to increase committed actions based on one's values.
- Wait-list Control Group: No intervention. This is a 'usual care' group.
Period: Overall Study
Arm/Group | Coping Effectiveness Training (CET) | Cognitive-behavioral Therapy (CBT) | Acceptance and Commitment Therapy | Wait-list Control Group
Started | 10 | 10 | 10 | 10
Completed | 6 | 4 | 7 | 8
Not Completed | 4 | 6 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coping Effectiveness Training (CET) | Cognitive-behavioral Therapy (CBT) | Acceptance and Commitment Therapy | Wait-list Control Group | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (18.9) | 56.9 (15.2) | 61.6 (17.6) | 60.7 (14.3) | 57.8 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 1 | 8
  Male | 9 | 8 | 6 | 9 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Coping
Description: The Brief COPE scale (Carver, 1997) is a widely-used 28-item short form of the COPE Inventory (Carver, Scheier et al., 1989). This instrument measures 14 coping subscales. Each item is scored using a 1-4 frequency scale (i.e., 1= "I haven't been doing this it at all" to 4= "I've been doing this a lot"), where higher scores reflect greater use of the coping strategy. A three-factor structure was used as follows: (a) Engagement coping (EC), including active coping, positive reframing, planning, accepting, and use of humor (items n = 12; score range 12-48); (b) disengagement coping (DC), including self-distancing, denial, behavioral disengagement, and self-blame (items n = 6; score range 6-24); and (c) social support coping (SS), including instrumenal support, emotional support, venting, and religion (items n = 8; score range 8-32).
Time Frame: Baseline
Population: Brief COPE 3 factors (engagement, disengagement, and social support)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coping Effectiveness Training (CET) | Cognitive-behavioral Therapy (CBT) | Acceptance and Commitment Therapy | Wait-list Control Group
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Engagement coping | 34.3 (1.2) | 31.6 (1.2) | 33.2 (1.2) | 30.0 (1.2)
  Disengagement coping | 9.6 (.6) | 7.4 (.6) | 8.7 (.6) | 7.6 (.6)
  Social support coping | 19.2 (.99) | 16.3 (.99) | 16.4 (.99) | 14.9 (.99)

ADVERSE EVENTS:
Time Frame: 2015-2016: one year of data collection.
Description: The Clinicaltrials.gov definition (i.e., "Any untoward or unfavorable medical occurrence in a participant...temporally associated with the participant's participation in the research...") was used. Given that the interventions were psychological, the data related to medical events were not collected by the research team; if any such medical events had been self-reported by participants, then the data will be reported to the Institutional Review Board and on the Clinicaltrials.gov website).
Arm/Group | Coping Effectiveness Training (CET) | Cognitive-behavioral Therapy (CBT) | Acceptance and Commitment Therapy | Wait-list Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
One limitation was that only self-report instruments were used, and therefore, social desirability may have influenced the results. Further, while this study involved repeated measures, the sample was small and thus the results should be replicated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes